CLINICAL TRIAL: NCT00104572
Title: The Effects of Aromatase Inhibition and Testosterone Replacement in Sex Steroids, Pituitary Hormones, Markers of Bone Turnover, Muscle Strength, and Cognition in Older Men
Brief Title: Effects of Aromatase Inhibition Versus Testosterone in Older Men With Low Testosterone: Randomized-Controlled Trial.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999904338; NCT00104572; 04-AG-N338 (Other: NIHCC)
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2016-03

CONDITIONS: Hypogonadism; Diabetes; Sarcopenia; Osteoporosis; Depression
Keywords: Estrogen; Glucose Tolerance; Bone Density; Quality-of-Life; Sarcopenia
MeSH Terms: conditions — Hypogonadism; Diabetes Mellitus; Sarcopenia; Osteoporosis; Depression | interventions — Testosterone; Anastrozole; Aromatase Inhibitors; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- (Androgel) testosterone gel (Experimental): 17 participants will receive testosterone gel (5 gm) plus placebo tablet daily for 12 months and 'Calcium Cardone 500mg with vitamin D 400 IU'
  Interventions: Drug: Androgel (Testosterone Gel); Drug: Placebo tablet; Dietary Supplement: Calcium Cardone 500mg with vitamin D 400 IU
- anastrozole (Aromatase inhibitor) (Experimental): 14 participants will receive anastrozole 1 mg tablet plus placebo gel daily for 12 months and 'Calcium Cardone 500mg with vitamin D 400 IU'
  Interventions: Drug: Anastrozole (Aromatase Inhibitor); Drug: Placebo gel; Dietary Supplement: Calcium Cardone 500mg with vitamin D 400 IU
- placebo (Placebo Comparator): 13 participants will receive a placebo tablet and placebo gel daily for 12 months and 'Calcium Cardone 500mg with vitamin D 400 IU'
  Interventions: Drug: Placebo tablet; Drug: Placebo gel; Dietary Supplement: Calcium Cardone 500mg with vitamin D 400 IU

INTERVENTIONS:
Drug: Androgel (Testosterone Gel) — 1 mg tablet for 12 months
  Arms: (Androgel) testosterone gel
Drug: Anastrozole (Aromatase Inhibitor)
  Arms: anastrozole (Aromatase inhibitor)
Drug: Placebo tablet — Daily for 12 months
  Arms: (Androgel) testosterone gel; placebo
Drug: Placebo gel — Daily for 12 months
  Arms: anastrozole (Aromatase inhibitor); placebo
Dietary Supplement: Calcium Cardone 500mg with vitamin D 400 IU — 1 tablet three times a day

SUMMARY:
Background: Men≥65 years often produce lower levels of testosterone, meaning there is less testosterone circulating to the tissues of the body. This is associated with negative effects on muscle strength, bone density, sexual function, mood, and the ability to think to the best of one's ability. Testosterone replacement therapy often involves injections, patches, or gels that help to raise circulating testosterone levels, but these therapies often have side effects because they lead to imbalance of other hormones. Researchers have been studying the effectiveness of anastrozole, a drug that can lower estrogen levels while simultaneously increasing testosterone levels, as a treatment for the negative effects of decreased circulating testosterone levels that occur naturally with aging. Objectives: To evaluate whether anastrozole is as effective as testosterone gel in improving bone and muscle strength, hormone levels, and brain function in men over 65 years of age. Eligibility: Healthy men at least 65 years of age who have low levels of testosterone. Design: The study involves six study visits over a total of 12 months: screening, baseline, 6 weeks, 3 months, 6 months, and 12 months. All participants will receive calcium and vitamin D supplements to take daily, and will be randomized to one of three groups:Testosterone gel and placebo tablet, Anastrozole tablet and placebo gel, Placebo tablet and gel. Participants will have the following tests at each specified visit:Screening: Blood tests and rectal ultrasound to evaluate the prostate;Baseline: Blood and urine tests; growth hormone levels, muscle strength, bone density, and balance evaluation; imaging studies; cognitive testing; and questionnaires on quality of life, sexual function, depression, and urinary symptoms;Six weeks: Blood tests and dose adjustment of the gel or tablet;Three months: Blood and urine tests; growth hormone, muscle strength, bone density, and balance evaluation; and questionnaires on quality of life, sexual function, depression, and urinary symptoms;Six months: Blood and urine tests; muscle strength, bone density, and balance evaluation; cognitive testing; and questionnaires on quality of life, sexual function, depression, and urinary symptoms;Twelve months: Blood and urine tests; rectal ultrasound; muscle strength, bone density, and balance evaluation; imaging studies; cognitive testing; and questionnaires on quality of life, sexual function, depression, and urinary symptoms.

DETAILED DESCRIPTION:
Approximately 20% of men over the age of 70 have low testosterone levels. In some studies, testosterone replacement has resulted in improvement in bone mass, muscle strength, quality of life and memory function. In the body, testosterone is converted into estrogen. Hence, it is unclear whether these beneficial effects are due to testosterone or estrogen. Research has shown that inhibition of estrogen production in men results in an increase in testosterone levels.

In this study, patients will be assigned to one of three groups: one group will receive testosterone gel and a placebo tablet, one group will receive a 1mg Anastrozole tablet and a placebo gel, and one group will receive a placebo tablet and placebo gel. Each group will receive a daily dose of calcium with vitamin D. The study requires 6 visits over a 12-month period for testing and evaluation. Two of the 6 visits will require an overnight stay in the hospital so that an intravenous (IV) line can be placed in the arm to allow samples to be drawn throughout the night. Testing will include a cardiac stress test, a glucose tolerance test, bone and muscle tests, evaluation of memory function, etc. For the safety of the prostate, we will perform a prostate ultrasound at the start and end of the study and we will monitor urinary symptoms, prostate specific antigen (PSA) levels and the prostate exam throughout the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Men age 65 years or older
  2. Serum testosterone level less than or equal to 350 ng/dl
  3. Subject is able to complete an informed consent

EXCLUSION CRITERIA:

1. History of Stroke
2. History of Dementia
3. History of Diabetes
4. Blood pressure at rest of > 155/90 mmHg. Elevated systolic or diastolic reading renders subject ineligible
5. Chronic medical condition, i.e. congestive heart failure
6. Arthritis, severe enough to prevent completion of the strength testing, history of joint replacement of knees or hip.
7. Inability to walk 50 meters
8. Known disease of the bone and/or taking medications to treat osteoporosis, i.e.

   Fosamax, Evista, Miacalcin
9. History of Gastric surgery
10. History of prostate cancer or any other cancers, including blood dyscrasias
11. History of severe benign prostatic hyperplasia (causing urinary problems)
12. History of heart attack or open-heart surgery within the past 6 months
13. Use of steroids within the past 3 months, including prednisone and/or cortisone injections, and inhaled steroids. Topical steroid cream is acceptable.
14. If you do not agree to refrain from taking the drugs Viagra, Cialis or Levitra for the duration of the study
15. Use of anabolic steroids, i.e. testosterone, (or any analog of testosterone) Dehydroepiandrosterone or any growth promoters i.e. growth hormone itself or analogs of growth hormone
16. Use of anti-androgen medications, i.e. Aldactone, Tagamet, Proscar, estrogens
17. Use of Dilantin or Phenobarbital
18. Alcohol intake > 30 grams (drink more than 2 beers per day OR more than 1 glass of wine or cocktail daily)
19. Currently smokes any tobacco product
20. Having started a new medication during the past three months which may interfere with the outcome measures of the study
21. Polycythemia
22. Prostate specific antigen > 4.0 ng/dl
23. Hematocrit < 36
24. Liver function tests greater than 2 times upper normal limits or abnormal electrolytes, calcium or Parathyroid hormone , at the discretion of the investigator
25. Mini Mental Status Exam score less than or equal to 24

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-03; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jeffcoate SL, Brooks RV, Lim NY, London DR, Prunty FT, Spathis GS. Androgen production in hypogonadal men. J Endocrinol. 1967 Apr;37(4):401-11. doi: 10.1677/joe.0.0370401. No abstract available. PMID 4290227
- [Background] Wheeler MJ. The determination of bio-available testosterone. Ann Clin Biochem. 1995 Jul;32 ( Pt 4):345-57. doi: 10.1177/000456329503200401. No abstract available. PMID 7486793
- [Background] Gray A, Feldman HA, McKinlay JB, Longcope C. Age, disease, and changing sex hormone levels in middle-aged men: results of the Massachusetts Male Aging Study. J Clin Endocrinol Metab. 1991 Nov;73(5):1016-25. doi: 10.1210/jcem-73-5-1016. PMID 1719016
- [Derived] Dias JP, Melvin D, Shardell M, Ferrucci L, Chia CW, Gharib M, Egan JM, Basaria S. Effects of Transdermal Testosterone Gel or an Aromatase Inhibitor on Prostate Volume in Older Men. J Clin Endocrinol Metab. 2016 Apr;101(4):1865-71. doi: 10.1210/jc.2016-1111. Epub 2016 Mar 7. PMID 26950683

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study randomized 44 subjects, however 9 of them stop the study before having the second visit completed, so we started the analysis with 35 subjects. The participant flow module has 35 subjects, because these subjects have a baseline and 3 months endpoints.
Groups:
- Transdermal Testosterone: 13 participants will receive testosterone gel (5 gm) plus placebo tablet daily for 12 months
  Androgel (Testosterone Gel): 1 mg tablet for 12 months
  Placebo tablet: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
- Aromatase Inhibitor: 13 participants will receive anastrozole 1 mg tablet plus placebo gel daily for 12 months
  Anastrozole (Aromatase Inhibitor)
  Placebo gel: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
- Placebo: 9 participants will receive a placebo tablet and placebo gel daily for 12 months
  Placebo tablet: Daily for 12 months
  Placebo gel: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
Period: Overall Study
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Started | 13 (These are the analysed subjects) | 13 (These are the analysed subjects) | 9 ((N=11) in placebo, physician removed 2 men due to total testosterone>450 ng/DL, N=9 analysed.)
Completed | 10 | 10 | 9
Not Completed | 3 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transdermal Testosterone: participants will receive testosterone gel (5 gm) plus placebo tablet daily for 12 months
  Androgel (Testosterone Gel): 1 mg tablet for 12 months
  Placebo tablet: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
- Aromatase Inhibitor: participants will receive anastrozole 1 mg tablet plus placebo gel daily for 12 months
  Anastrozole (Aromatase Inhibitor)
  Placebo gel: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
- Placebo: participants will receive a placebo tablet and placebo gel daily for 12 months
  Placebo tablet: Daily for 12 months
  Placebo gel: Daily for 12 months
  Calcium Cardone 500mg with vitamin D 400 IU: 1 tablet three times a day
- Total: Total of all reporting groups
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (5.1) | 70 (3.0) | 72 (3.4) | 71 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 13 | 9 | 35
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 9 | 35
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.8 (9.4) | 134.5 (14.5) | 133.7 (11.2) | 135.3 (2.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 73.3 (5.3) | 72.4 (9.4) | 73.1 (10.4) | 72.9 (0.5)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 30.1 (4.0) | 27.8 (4.1) | 27.6 (3.5) | 28.5 (1.4)
Total Testosterone [Mean (Standard Deviation); unit: ng/dL] | 300.1 (81.9) | 271.6 (85.6) | 303.8 (94.7) | 291.8 (17.6)
Bioavailable Testosterone [Mean (Standard Deviation); unit: ng/dL] | 114.4 (37.2) | 114.8 (36.3) | 91.2 (31.7) | 106.8 (13.5)
Estradiol [Mean (Standard Deviation); unit: ng/dL] | 2.0 (0.7) | 1.5 (0.6) | 1.6 (0.5) | 1.700 (0.3)
Sex hormone-binding globulin [Mean (Standard Deviation); unit: nmol/L] | 43.4 (22.2) | 39.9 (19.4) | 58.6 (21.3) | 47.30 (10.0)
luteinizing hormone [Mean (Standard Deviation); unit: mlU/ml] | 11.4 (8.2) | 6.4 (2.7) | 12.2 (10.1) | 10.00 (3.1)
follicle-stimulating hormone [Mean (Standard Deviation); unit: mlU/ml] | 8.0 (6.4) | 6.5 (5.3) | 8.2 (10.9) | 7.567 (0.9)
Bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 1.4 (0.2) | 1.3 (0.2) | 1.2 (0.1) | 1.3 (0.1)
lean body mass [Mean (Standard Deviation); unit: kg] | 56.0 (12) | 54.7 (11.0) | 56.0 (7.2) | 55.6 (0.8)
Fat mass [Mean (Standard Deviation); unit: kg] | 31.6 (10.4) | 26.9 (9.6) | 28.5 (7.6) | 29.0 (2.4)
hand grip [Mean (Standard Deviation); unit: kg] | 41.1 (6.9) | 39.2 (9.9) | 39.3 (7.2) | 39.9 (1.1)
knee strength [Mean (Standard Deviation); unit: Nm] | 133.8 (44.3) | 138.7 (48.6) | 155.4 (41.9) | 142.6 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Testosterone Gel vs. Anastrozole on Bone Mineral Density
Description: bone mineral density lumbar spine for all arms testosterone gel, anastrozole and placebo
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Number analyzed (Participants) | 13 | 13 | 9
g/cm2 | 0.042 (0.008) | 0.008 (0.012) | 0.047 (0.013)

2. Secondary Outcome: Effect of Testosterone Gel vs. Anastrozole on Pulsatile Growth Hormone Release
Description: Overnight Growth hormone measures (total hormone secretion) for groups testosterone gel, anastrozole and placebo
Time Frame: 1 year
Measure: Mean (Standard Error); unit: ng/ml/8h
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Number analyzed (Participants) | 13 | 13 | 9
ng/ml/8h | 5.8 (1.4) | 10 (2.2) | 7.7 (2.2)

3. Secondary Outcome: Effect of Testosterone Gel vs. Anastrozole on Glucose Tolerance/Lipid Metabolism
Description: Primary outcome HOMA-IR for all groups testosterone gel, anastrozole and placebo Insulin resistance measure by HOMA-IR is a score if a person is insulin resistance the score should be between minimum 0.7- maximum 2 or more.
  Absolute changes in HOMAIR in all treatment arms, calculation time frame 1 year minus baseline point.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Number analyzed (Participants) | 10 | 10 | 9
score on a scale | -0.05 (0.21) | 0.15 (0.10) | -0.11 (0.26)

4. Secondary Outcome: Effect of Testosterone Gel vs. Anastrozole on Prostate Volume/Prostate Specific Antigen Levels/Urinary Function
Description: rectal ultrasound prostate volume for all groups testosterone gel, anastrozole and placebo.
  Absolute changes in prostate volume in all treatment arms, calculation time frame 1 year minus baseline point.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: cc
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Number analyzed (Participants) | 10 | 10 | 9
cc | 4.5 (1.76) | -1.66 (3.54) | -1.05 (1.52)

ADVERSE EVENTS:
Description: The study randomized 44 subjects, however 9 of them stop the study before having the second visit completed, so we started the analysis with 35 subjects. The participant flow module has 35 subjects, because these subjects have a baseline and 3 months endpoints.
Arm/Group | Transdermal Testosterone | Aromatase Inhibitor | Placebo
Serious Adverse Events (participants affected / at risk) | 3/17 | 6/14 | 3/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Testosterone (N=17) | Aromatase Inhibitor (N=14) | Placebo (N=13)
muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — in aromatase group
bladder mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — bladder mass on transrectal exam
subdural hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
stent placement (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
mildly elevated HCT (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
elevated PSA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
increased heart rate palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
dizziness/diarrhea (General disorders) | 0 (0) | 1 (1) | 0 (0)
elevated PSA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
blood in semen (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes